CLINICAL TRIAL: NCT06869005
Title: Prévoir Les NAusées Et Vomissements CHimio Ou Radio-induits Chez Les Enfants/adolescents Traités Pour Un Cancer
Brief Title: Predict CHimio-or Radiation-induced NAusea and Vomiting in Children/adolescents Treated for Cancer
Acronym: PaNACHE
Status: Not yet recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC21_9789_PaNACHE
Record Dates: First submitted 2024-06-19; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Childhood Cancer; Nausea with Vomiting Chemotherapy-Induced
Keywords: Childhood Cancer; Chemo- or Radiation-induced Nausea and Vomiting (CVRN),; BARF scale; PaNACHE score
MeSH Terms: conditions — Neoplasms; Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: BARF scale — BARF Scale, validated in paediatrics, is graduated from 0 to 10 and shows 6 increasingly nauseous faces. A child/adolescent will be considered "at risk of NV" if he/she declares a score greater than or equal to 4 out of 10 on at least one of the 4 observation times.
  This scale can be used by the child him/herself, from the age of 4; or by a close adult, usually present at the child's side during treatment.

SUMMARY:
Chemo- or radiation-induced nausea and vomiting (CRVN) is one of the most frequent and feared side effects.

It is a symptom that is few or not at all evaluated. There is a significant discrepancy between the perception of the CRVN symptom by caregivers and the patient's own experience.

At present, there is no real consensus to manage CRVN with medication, and CRVN relief is also the subject of heterogeneous practices. The importance of primary prevention of CRVN, before starting the first treatment sequence, has been highlighted to optimize the action of antiemetic treatments and limit the risk of anticipated nausea and vomiting (NV).

The investigators' objective is to objectively assess the risk of CRVN in children/adolescents treated for cancer (and thus effectively prevent this symptom).

DETAILED DESCRIPTION:
In France, around 2,500 cancers are diagnosed each year in children/adolescents (0-18 years) (INCa data for 2011-2014).

For around 90% of these cases, chemotherapy and/or radiotherapy are indicated. Today, pediatric onco-hematology teams are committed to both the efficacy of treatments (and continue the progress made over the last few the progress made in recent decades in terms of survival); and to optimize the quality of life. One of the key areas for improving patient experience is to reduce the toxicity of treatments, and to prevent and alleviate known side effects.

Among these toxicities, chemo- or radiation-induced nausea and vomiting (CRVN) are one of the most frequent and dreaded side effects.

In addition to the impact of nausea and vomiting (NV) on the quality of life of children/adolescents (possibly impacting therapeutic); CRVN can lead to serious metabolic complications (sometimes impacting optimal treatment).

Theoretical considerations:

Several publications have already described the mechanisms of CRVN. Various studies have highlighted individual factors (gender, age, etc.) influencing the occurrence of NV (including in children/adolescents); and a variable emetogenic potential depending on the type of chemotherapy or radiotherapy.

- Several studies have focused on the prevention and relief of CVRN, a major side effect of cancer treatment. The importance of primary prevention of CVRN, before starting the first treatment sequence, has been highlighted.

The interests are twofold: to optimize the action of antiemetic treatments (more effective preventively than after the onset of vomiting); and to limit the risk of anticipated NV during subsequent treatment sequences.

- Finally, several observations made in different pediatric oncohaematology units, have highlighted a significant discrepancy between caregivers' perception of the CVRN symptom and the patient's own experience. These studies also highlight the existence of NV assessment scales, validated in pediatrics, but little known by professionals and therefore rarely used.

In practice:

* Currently, in pediatric onco-hematology, there is no real management of CVRN. Each team refers to a "local" procedure, and its application is often "left" to the discretion of each caregiver (prescription "if necessary"). A review of practices and therapeutic recommendations of the Support Care Committee of the SFCE (Société Française de lutte contre les Cancers et Leucémies des Enfants et adolescents) have recently been published.
* Relief of CVRN using non-medicinal techniques (hypnosis, acupuncture, laser, aromatherapy...) is also a heterogeneous practice (depending on specific professional skills), not evaluated in pediatrics.

In this context, the investigators were interested in the primary prophylaxis of NV; and wondered how to objectively assess the risk of CVRN in children/adolescents treated for cancer (and thus effectively prevent this symptom).

To meet this need, the project aims to develop a multifactorial score for assessing the risk of CVRN in children/adolescents treated for cancer (PaNACHE score).

The questioning at the origin of this project focused on considering the "NV" symptom in its different dimensions (sensory- emotional-cognitive-behavioral), such as the "pain" symptom. This approach enables us to base on validated models for assessing and managing pain in children/adolescents, centered in particular on the self-assessment of "patient experience".

The PaNACHE score is based on :

Assessment of various factors (individual and/or treatment-related) influencing NV (some of which have already been described in the literature)

- Self-assessment of NV perceived by the children/adolescent using the BARF scale (BAxter Retching Faces). This scale, graded from 0 to 10, shows 6 increasingly nauseous faces. It has been validated in pediatrics.

It can be used by the child himself from the age of 4, or by a close adult who is usually present with the child during treatment.

Since several studies have highlighted a noticeable difference between the caregiver's perception of the CVRN symptom and the patient's own experience, the investigators feel it is important to take into account the child/adolescent's self-assessment of his or her feelings, and not simply the factual number of vomits and/or the caregiver's hetero-assessment of perceived nausea.

ELIGIBILITY:
Inclusion Criteria:

* Treated in a pediatric onco-hematology center in the GOCE (Grand Ouest Cancer Enfant) inter-region;
* Receiving chemotherapy or radiotherapy;
* According to patient age :
* Minor (under 18 years): At least one parent has been informed of the protocol and has not expressed opposition to the child's participation in the study
* Adult (more than 18 years): Having received information about the protocol and not having expressed opposition to participating in the study

Exclusion Criteria:

* Patients or legal representatives with French understanding difficulties.
* Patients or legal representatives subject with legal protection (safeguard of justice, curatorship, guardianship) or deprived of liberty.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In the Grand Ouest region, around 400 children/adolescents (aged 0-18) are diagnosed with cancer every year.
  A sample of 150 subjects is expected for this research (involving 5 of the 10 GOCE collaborating centers).
  This sample will be used to create a score including around ten variables (Peduzzi 1995).
  The distribution of the number of inclusions is adapted to the recruitment and activity (chemotherapy or radiotherapy) of each of the 5 centers participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Develop a multifactorial score to evaluate the risk of CVRN in children/adolescents treated for cancer (PaNACHE score). | Up to 6 weeks.
  The primary outcome is a score based on :
  * Dependent variable, binary, corresponding to self-assessment of NV perceived by the child/adolescent with the BARF Scale. This scale, validated in pediatrics, is graduated from 0 to 10 and shows 6 faces of increasing nausea. A child/adolescent will be considered "at risk of NV" if they report a score greater than or equal to 4 out of 10 on at least one of the 4 observation times.
  * Predictive variables, likely to influence NV: Individual variables (age, sex, history of NV, etc.) and treatment-related variables (type of chemotherapy, area and dose of irradiation).

SECONDARY OUTCOMES:
Evaluate the concordance between the hetero-assessment of NV perceived by caregivers and the self-assessment of NV experienced by the patient. | Up to 6 weeks.
  In order to objectify professional practices, the child/adolescent's self-assessment of perceived NV (via the BARF Scale) will be compared with the caregiver's hetero-assessment (via the same BARF Scale) compared with caregiver hetero-assessment (using the same BARF Scale).
Describe the management methods (preventive and/or curative; medicinal and/or non-medicinal) for CRVN, throughout the treatment phase. | Up to 6 weeks.
  Management methods (preventive and/or curative; medication and/or non-medication) for CRVN will be recorded for each patient, at each of the 4 observation times specified in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Maïna LETORT-BERTRAND, Principal Investigator — CHU Rennes Hôpital Sud
Locations (5):
- France (5):
  - CHU Angers, Angers, France
  - CHU Caen FEH, Caen, France
  - Rennes University Hospital, Rennes, France
  - Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain, France
  - CHU Tours Hôpital Clocheville, Tours, France

IPD SHARING:
Plan to Share IPD: No